CLINICAL TRIAL: NCT03834662
Title: A Phase 1 Cohort Dose-Escalation Trial of AVID200, a Transforming Growth Factor β (TGFβ) Inhibitor, in Patients With Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Trial of AVID200, a Transforming Growth Factor β (TGFβ) Inhibitor, in Patients Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Formation Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVID200-03
Record Dates: First submitted 2019-01-31; First posted 2019-02-08 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Malignant Solid Tumor
Keywords: Solid tumors

STUDY DESIGN:
Intervention Model Description: Evaluation of the safety, tolerability, and dose-limiting toxicities (DLTs), to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of sequential escalating doses of AVID200 when administered once every 3 weeks (Q3W) by IV infusion to patient cohorts (3)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1: 180 mg/m2 of AVID200 (Experimental): Intravenous infusion of AVID200 over 1 hour administered every three weeks. Starting dose for dose escalation.
  Interventions: Drug: AVID200
- Dose Level 2: 550 mg/m2 of AVID200 (Experimental): Intravenous infusion of AVID200 over 1 hour administered every three weeks.
  Interventions: Drug: AVID200
- Dose Level 3: 1100 mg/m2 (Experimental): Intravenous infusion of AVID200 over 1.5 hours administered every three weeks.
  Interventions: Drug: AVID200

INTERVENTIONS:
Drug: AVID200 — A TGFβ receptor ectodomain-IgG Fc fusion protein inhibitor of TGFβ
  Other Names: TGFβ receptor ectodomain-IgG Fc fusion protein

SUMMARY:
TGFβ has profound local immunosuppressive and immunoexclusion effects in the tumor microenvironment that are integrally involved in the failure of immune checkpoint inhibitors in some tumors. Preclinical data in a variety of models strongly support the study of AVID200 in patients with treatment-refractory advanced and metastatic malignancies as an approach to reducing immunosuppression/exclusion and increasing the activity of immune checkpoint inhibitors.

DETAILED DESCRIPTION:
TGFβ inhibits local anti-tumor immunity in the tumor microenvironment (TME) and also promotes the epithelial to mesenchymal transition (EMT) that enhances the metastatic potential of tumor cells. Cancer-associated fibroblasts (CAFs) are a critical constituent of the TME. As is the case for fibrosis in other settings, these cells are myofibroblast-like, and respond to and are activated by tumor-derived TGFβ. CAFs play a critical role in promoting EMT resulting in increased tumor cell migration and invasion as well as maintaining the TME to support tumor cell survival. The immunosuppressive role of TGFβ in the TME has been clearly demonstrated with the activation of CAFs being an important mechanism underlying immune cell exclusion. Exclusion of immune cells from tumors and local immunosuppression can both be reversed by AVID200 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented (histologically or cytologically proven) solid tumor malignancy that is locally advanced or metastatic
* Patients with a malignancy that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor
* Patients with a malignancy that is either refractory to, or the patient is intolerant of existing therapy(ies) known to provide clinical benefit, or for which no standard therapy is available
* Patients with measurable or non-measurable disease according to RECIST, v1.1
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (or equivalent Karnofsky PS), and anticipated life expectancy of ≥ 3 months
* Patients and their partners who are either not of childbearing potential or who agree to use a highly effective, non-hormonal, method of contraception during the study and continuing until 4 months after the last dose of study drug); male patients agreeing to refrain from sperm donation during this period.
* Patients with the ability to understand and give written informed consent for participation

Exclusion Criteria:

* Patients with an active second malignancy or history of another malignancy within the last 2 years with the exception of:

  * Treated non-melanoma skin cancers
  * Treated carcinoma in situ (CIS) of the breast, cervix, bladder, colon, endometrium, skin (melanoma) provided complete response (CR) was achieved at least 2 years prior to study and no additional therapy is ongoing or required during study period with the exception of anti-estrogen/androgen therapy or bisphosphonates
  * Controlled, superficial carcinoma of the bladder
  * T1a carcinoma of the prostate comprising < 5% of resected tissue and prostate specific antigen (PSA) within normal limits (WNL) since resection
* Any antineoplastic agent for the primary malignancy (standard or investigational), without delayed toxicity, within 4 weeks or 5 plasma half-lives, whichever is shortest, prior to C1/D1 and during study with the exception of:

  -Nitrosoureas and mitomycin C within 6 weeks prior to C1/D1 and during study
* Any other investigational treatments within 4 weeks prior to and during study; includes participation in any medical device or supportive care therapeutic intervention trials
* Radiotherapy for target lesions within 4 weeks prior to C1/D1 and during study; radiotherapy for non-target lesions within 2 weeks prior to C1/D1
* Radiotherapy within 2 weeks prior to C1/D1 and during study. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Use of live vaccines against infectious diseases 4 weeks prior to C1/D1 and during study
* Immunosuppressive or systemic hormonal therapy (> 10 mg daily prednisone or equivalent) within 2 weeks prior to C1/D1 and during study
* Prophylactic use of hematopoietic growth factors within 2 weeks prior to C1/D1 and during Cycle 1 of study; thereafter prophylactic use of growth factors is allowed as clinically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, for up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Paul I Nadler, MD, Study Director — Forbius (Formation Biologics)
Locations (3):
- United States (2):
  - START Midwest Clinic, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No